CLINICAL TRIAL: NCT05316415
Title: The Effects of Music on the Anxiety and Sleep Quality of Pregnant Women on Bed Rest for a High-risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cemile Onat Koroglu, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017/65
Record Dates: First submitted 2022-02-14; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy, High Risk; Anxiety State; Sleep Quality
Keywords: Anxiety; bed rest; high-risk pregnancy; music; sleep quality
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acemaşiran Music Group (Experimental): Listening to Acemaşiran music for 40 minutes in successive three days and two times a day (noon and evening) Routine clinical care
  Interventions: Other: Acemaşiran Music Group
- Control Group (No Intervention): Routine clinical care

INTERVENTIONS:
Other: Acemaşiran Music Group — Agreeing to participate in the study Knowing Turkish and being literate Having been hospitalized for bed rest for at least 5 days. Having a gestational age of 28 to 36 weeks Being hospitalized due to at least one of the diagnoses including hypertensive diseases, diabetes mellitus, preterm labor, placenta previa, cervical insufficiency, or premature rupture of the membrane
  Arms: Acemaşiran Music Group

SUMMARY:
The purpose of this study is to identify the effects of music on the anxiety and sleep quality of women with high-risk pregnancy having bed rest in the hospital in Turkey.

This randomized-controlled study involved 80 control and 80 experimental group with a high-risk pregnant woman .

DETAILED DESCRIPTION:
The literature review indicates a limited number of studies on the effects of music in eliminating the anxiety and sleep problems in women with a high-risk pregnancy having bed rest in the hospital; the existing studies were found to be mainly about anxiety. The purpose of this study is to identify the effects of music on the anxiety and sleep quality of women with a high-risk pregnancy having bed rest in the hospital.

This study adopted a pretest-posttest randomized controlled study involved 80 control and 80 experimental group with a high-risk pregnant woman . The women in the experimental group listened to Acemaşiran music for 40 minutes in successive three days and two times a day.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Knowing Turkish and being literate
* Having been hospitalized for bed rest for at least 5 days.
* Having a gestational age of 28 to 36 weeks
* Being hospitalized due to at least one of the diagnoses including hypertensive diseases, diabetes mellitus, preterm labor, placenta previa, cervical insufficiency, or premature rupture of the membrane

Exclusion Criteria:

* Fetal congenital anomalies
* Having a hearing impairment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
State-trait Anxiety Inventory | Two hours after the last listening session, the participants were administered the State-trait anxiety inventory to measure
  The inventory developed by Spielberger et al. in 1970 consists of two parts that measure two different aspects of anxiety, which are state and trait anxiety. Two inventories are printed on separate pages, and each inventory has 20 questions

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | . Two hours after the last listening session, the participants were administered the Pittsburg Sleep Quality Index to measure their sleep quality.
  The PSQI consists of 19 self-rated questions, and 5 questions rated by the bedpartner or roommate. The 19 self-rated questions assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep-related problems. Each subscale is scored between 0 and 3, and the total score to be obtained from the scale ranges between 0 and 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University Balcalı Hospital, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No